CLINICAL TRIAL: NCT01384578
Title: A Randomized Controlled Project to Study the Efficacy of Combined Pentoxiphylline and Vitamin E Versus Vitamin E in Patients With Non- Alcoholic Steatohepatitis
Brief Title: Pentoxiphylline and Vitamin E Versus Vitamin E in Patients With Non- Alcoholic Steatohepatitis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of funds
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-NASH-02
Record Dates: First submitted 2011-06-28; First posted 2011-06-29 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2012-07

CONDITIONS: Non Alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- pentoxiphylline and Vitamin E (Experimental)
  Interventions: Drug: pentoxiphylline and Vitamin E
- Vitamin E (Active Comparator)
  Interventions: Drug: Vitamin E

INTERVENTIONS:
Drug: pentoxiphylline and Vitamin E — Patients in cases group (Group 1) will receive pentoxiphylline (PTX) 400 mg thrice daily and vitamin E 800 IU/day.
  Arms: pentoxiphylline and Vitamin E
Drug: Vitamin E — Patients in control group will receive vitamin E 800 IU/day
  Arms: Vitamin E

SUMMARY:
120 patients of biopsy proven NASH will be randomized into two groups. Cases group will receive combination of pentoxiphylline and Vitamin E, and control group will receive only Vitamin E.

DETAILED DESCRIPTION:
The investigators plan to randomise 120 patients of biopsy proven NASH into cases and control groups.

Baseline investigations:

Clinical characteristics

* Age
* Gender
* Anthropometry (BMI, waist circumference, waist- hip ratio, triceps skin fold thickness, mid arm circumference)
* Alcohol intake should be nil

Laboratory characteristics

* Hemogram, INR, KFT
* LFT (especially ALT, GGT) , APRI (AST to platelet ratio)
* Fasting Lipid Profile
* Other possible etiologies of liver disease (viral markers, ferritin, ANA, IgG, ceruloplasmin )
* HOMA-IR (II)
* Serum uric acid levels Liver stiffness
* Fibroscan
* MR elastography Radiological characteristics
* USG abdomen Variceal status by UGI endoscopy Alpha fetoprotein Pro- inflammatory markers
* TNF-alpha, IL-6, adiponectin, leptin and osteopontin Liver biopsy and NAS score

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years
* Persistently abnormal ALT >1.2 times upper limit of normal
* Histological evidence of NASH/cirrhosis on liver biopsy. ( The minimal criteria for diagnosis of NASH included the presence of lobular inflammation and either ballooning of cells or perisinusoidal or pericellular fibrosis in Zone 3 of the hepatic acinus)

Exclusion Criteria:

* A known case of Type 2 diabetes mellitus on treatment
* Alcohol intake of more than 40gm / week
* If they had evidence of cirrhosis with significant portal hypertension
* Ongoing total parenteral nutrition/ jejunal-ileal bypass
* Other known liver disease (Hepatitis A to E, autoimmune liver disease, Wilson's disease, alpha 1 antitrypsin deficiency and hemochromatosis)
* Medication like estrogens, amiodarone, MTx, tamoxifen, ATT
* Pregnancy or lactation
* Hypersensitivity to methylxanthines (e.g., caffeine, theophylline, theobromine )
* Recent retinal/cerebral hemorrhage
* Acute myocardial infarction or severe cardiac arrhythmias
* Impaired renal function
* Hypothyroidism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
histological outcome in the form of improvement or non- progression in hepatocyte injury and fibrosis (NAS score). | 3 Months

SECONDARY OUTCOMES:
Response in form of anthropometry , HOMA-IR, fasting lipid profiles, biochemical response in form of normalization of ALT and AST levels and reduction in uric | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Shiv Kumar Sarin, MD,DM, Study Director — Institute of Liver & Biliary Sciences (ILBS)
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Kedarisetty CK, Bhardwaj A, Kumar G, Rastogi A, Bihari C, Kumar M, Sarin SK. Efficacy of combining pentoxiphylline and vitamin E versus vitamin E alone in non-alcoholic steatohepatitis- A randomized pilot study. Indian J Gastroenterol. 2021 Feb;40(1):41-49. doi: 10.1007/s12664-020-01131-x. Epub 2021 Mar 27. PMID 33772456